CLINICAL TRIAL: NCT05238831
Title: Serial Measurements of Molecular and Architectural Responses to Therapy (SMMART) Trial: Adaptive Clinical Treatment (ACT)
Brief Title: SMMART Adaptive Clinical Treatment (ACT) Trial
Status: Withdrawn | Phase: Early Phase 1 | Type: Interventional
Why Stopped: Withdrawn due to a change in therapeutic interventions.
Sponsor: OHSU Knight Cancer Institute (Other)
Collaborators: Genentech, Inc. (Industry); Oregon Health and Science University (Other)
Responsible Party: Principal Investigator, Lara Davis, MD, Principal Investigator, OHSU Knight Cancer Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: STUDY00020679; NCI-2021-12938 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); STUDY00020679 (Other: OHSU Knight Cancer Institute)
Record Dates: First submitted 2022-02-09; First posted 2022-02-14 (Actual); Last update posted 2024-01-23 (Actual); Status verified 2024-01

CONDITIONS: Advanced Breast Carcinoma; Advanced Malignant Solid Neoplasm; Advanced Ovarian Carcinoma; Advanced Pancreatic Carcinoma; Advanced Prostate Carcinoma; Advanced Sarcoma; Anatomic Stage III Breast Cancer AJCC v8; Anatomic Stage IV Breast Cancer AJCC v8; Recurrent Adult Soft Tissue Sarcoma; Recurrent Breast Carcinoma; Recurrent Ovarian Carcinoma; Recurrent Prostate Carcinoma; Stage II Pancreatic Cancer AJCC v8; Stage III Ovarian Cancer AJCC v8; Stage III Pancreatic Cancer AJCC v8; Stage IV Ovarian Cancer AJCC v8; Stage IV Pancreatic Cancer AJCC v8
MeSH Terms: conditions — Sarcoma; Breast Neoplasms; Ovarian Neoplasms; Prostatic Neoplasms; Pancreatic Neoplasms | interventions — alectinib; Alpelisib; Anastrozole; atezolizumab; Bevacizumab; Immunoglobulin G; Disulfides; Biopsy; Specimen Handling; Capecitabine; Carboplatin; cobimetinib; entrectinib; eribulin; Fulvestrant; Trastuzumab; pertuzumab; Irinotecan; Letrozole; 130-nm albumin-bound paclitaxel; Albumin-Bound Paclitaxel; Taxes; niraparib; olaparib; Paclitaxel; palbociclib; 2C4 antibody; PF-05280014; Ogivri; Ontruzant; trastuzumab biosimilar HLX02; Ado-Trastuzumab Emtansine; Vemurafenib; Vinorelbine; HhAntag691

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (SMMART-ACT) (Experimental): Administered in monotherapy or in combination with other targeted agents or immunotherapies, chemotherapies, or radiation. Combination treatment plans may include a two-week monotherapy lead-in, followed by a combination treatment regimen. Each ACT study intervention must have an established RP2D determined in a prior clinical trial. Participants undergo a Pre-Treatment Biopsy, plus an On-Treatment Biopsy after two weeks on first dose of study drug(s) and prior to starting Cycle 2, regardless of regimen. Participants continue to receive study agent(s) after the On-Treatment Biopsy, according to the biopsy results and the results of ongoing safety and clinical assessments. Treatment cycles repeat every 21 to 28 days in the absence of disease progression or unacceptable toxicity. Cycles are determined based on the study agent(s). Upon disease progression, participants are given the option to undergo an additional biopsy.
  Interventions: Drug: Alectinib; Drug: Alpelisib; Drug: Anastrozole; Biological: Atezolizumab; Biological: Bevacizumab; Procedure: Biopsy; Procedure: Biospecimen Collection; Drug: Capecitabine; Drug: Carboplatin; Drug: Cobimetinib; Drug: Entrectinib; Drug: Eribulin; Drug: Fulvestrant; Biological: Hyaluronidase-zzxf/Pertuzumab/Trastuzumab; Drug: Irinotecan; Drug: Letrozole; Drug: Nab-paclitaxel; Drug: Niraparib; Drug: Olaparib; Drug: Paclitaxel; Drug: Palbociclib; Biological: Pertuzumab; Other: Quality-of-Life Assessment; Biological: Trastuzumab; Biological: Trastuzumab Emtansine; Drug: Vemurafenib; Drug: Vinorelbine; Drug: Vismodegib

INTERVENTIONS:
Drug: Alectinib — Given orally (PO)
  Other Names: AF-802; AF802; Alecensa; ALK Inhibitor RO5424802; CH5424802; RG7853; RO5424802
Drug: Alpelisib — Given PO
  Other Names: BYL719; Phosphoinositide 3-kinase Inhibitor BYL719; Piqray; VIJOICE
Drug: Anastrozole — Given PO
  Other Names: Anastrazole; Arimidex; ICI D1033; ICI-D1033; ZD-1033
Biological: Atezolizumab — Given IV
  Other Names: MPDL 3280A; MPDL 328OA; MPDL-3280A; MPDL3280A; MPDL328OA; RG7446; RO5541267; Tecentriq
Biological: Bevacizumab — Given IV
  Other Names: ABP 215; Anti-VEGF; Anti-VEGF Humanized Monoclonal Antibody; Anti-VEGF Monoclonal Antibody SIBP04; Anti-VEGF rhuMAb; Avastin; Bevacizumab awwb; Bevacizumab Biosimilar ABP 215; Bevacizumab Biosimilar BEVZ92; Bevacizumab Biosimilar BI 695502; Bevacizumab Biosimilar CBT 124; Bevacizumab Biosimilar CT-P16; Bevacizumab Biosimilar FKB238; Bevacizumab Biosimilar GB-222; Bevacizumab Biosimilar HD204; Bevacizumab Biosimilar HLX04; Bevacizumab Biosimilar IBI305; Bevacizumab Biosimilar LY01008; Bevacizumab Biosimilar MIL60; Bevacizumab Biosimilar Mvasi; Bevacizumab Biosimilar MYL-1402O; Bevacizumab Biosimilar QL 1101; Bevacizumab Biosimilar QL1101; Bevacizumab Biosimilar RPH-001; Bevacizumab Biosimilar SCT501; Bevacizumab Biosimilar Zirabev; Bevacizumab-awwb; Bevacizumab-bvzr; BP102; BP102 Biosimilar; HD204; Immunoglobulin G1 (Human-Mouse Monoclonal rhuMab-VEGF Gamma-Chain Anti-Human Vascular Endothelial Growth Factor), Disulfide With Human-Mouse Monoclonal rhuMab-VEGF Light Chain, Dimer; Mvasi; MYL-1402O; QL1101; Recombinant Humanized Anti-VEGF Monoclonal Antibody; rhuMab-VEGF; SCT501; SIBP 04; SIBP-04; SIBP04; Zirabev
Procedure: Biopsy — Undergo tissue biopsy
  Other Names: BIOPSY_TYPE; Bx
Procedure: Biospecimen Collection — Undergo collection of blood
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Drug: Capecitabine — Given PO
  Other Names: Ro 09-1978/000; Xeloda
Drug: Carboplatin — Given IV
  Other Names: Blastocarb; Carboplat; Carboplatin Hexal; Carboplatino; Carboplatinum; Carbosin; Carbosol; Carbotec; CBDCA; Displata; Ercar; JM-8; Nealorin; Novoplatinum; Paraplatin; Paraplatin AQ; Paraplatine; Platinwas; Ribocarbo
Drug: Cobimetinib — Given PO
  Other Names: Cotellic; GDC-0973; MEK Inhibitor GDC-0973; XL518
Drug: Entrectinib — Given PO
  Other Names: Rozlytrek; RXDX 101; RXDX-101; RXDX101
Drug: Eribulin — Given IV
  Other Names: ER-086526
Drug: Fulvestrant — Given by injection
  Other Names: Faslodex; Faslodex(ICI 182,780); ICI 182,780; ICI 182780; ZD9238
Biological: Hyaluronidase-zzxf/Pertuzumab/Trastuzumab — Given phesgo SC
  Other Names: Pertuzumab, Trastuzumab, and Hyaluronidase-zzxf; Pertuzumab/Trastuzumab/Hyaluronidase-zzxf; Phesgo
Drug: Irinotecan — Given IV
Drug: Letrozole — Given PO
  Other Names: CGS 20267; Femara
Drug: Nab-paclitaxel — Given IV
  Other Names: ABI 007; ABI-007; Abraxane; Albumin-bound Paclitaxel; Albumin-Stabilized Nanoparticle Paclitaxel; Nanoparticle Albumin-bound Paclitaxel; Nanoparticle Paclitaxel; Paclitaxel Albumin; paclitaxel albumin-stabilized nanoparticle formulation; Protein-bound Paclitaxel
Drug: Niraparib — Given PO
  Other Names: MK-4827; MK4827
Drug: Olaparib — Given PO
  Other Names: AZD 2281; AZD-2281; AZD2281; KU-0059436; Lynparza; PARP Inhibitor AZD2281
Drug: Paclitaxel — Given IV
  Other Names: Anzatax; Asotax; Bristaxol; Praxel; Taxol; Taxol Konzentrat
Drug: Palbociclib — Given IV
  Other Names: 6-Acetyl-8-cyclopentyl-5-methyl-2-((5-(piperazin-1-yl)pyridin-2-yl)amino)-8h-pyrido(2,3-d)pyrimidin-7-one; Ibrance; PD 0332991; PD 332991; PD 991; PD-0332991
Biological: Pertuzumab — Given subcutaneously (SC)
  Other Names: 2C4; 2C4 Antibody; EG1206A; HLX11; HS627; MoAb 2C4; Monoclonal Antibody 2C4; Omnitarg; Perjeta; Pertuzumab Biosimilar EG1206A; Pertuzumab Biosimilar HLX11; Pertuzumab Biosimilar HS627; rhuMAb2C4; RO4368451
Other: Quality-of-Life Assessment — Ancillary studies
  Other Names: Quality of Life Assessment
Biological: Trastuzumab — Given SC
  Other Names: ABP 980; ALT02; Anti-c-ERB-2; Anti-c-erbB2 Monoclonal Antibody; Anti-ERB-2; Anti-erbB-2; Anti-erbB2 Monoclonal Antibody; Anti-HER2/c-erbB2 Monoclonal Antibody; Anti-p185-HER2; c-erb-2 Monoclonal Antibody; HER2 Monoclonal Antibody; Herceptin; Herceptin Biosimilar PF-05280014; Herceptin Trastuzumab Biosimilar PF-05280014; Herzuma; Kanjinti; MoAb HER2; Monoclonal Antibody c-erb-2; Monoclonal Antibody HER2; Ogivri; Ontruzant; PF-05280014; QL 1701; QL-1701; QL1701; rhuMAb HER2; RO0452317; SB3; Trastuzumab Biosimilar ABP 980; Trastuzumab Biosimilar ALT02; trastuzumab biosimilar EG12014; Trastuzumab Biosimilar HLX02; Trastuzumab Biosimilar PF-05280014; Trastuzumab Biosimilar QL1701; Trastuzumab Biosimilar SB3; Trastuzumab Biosimilar SIBP-01; Trastuzumab-anns; Trastuzumab-dkst; Trastuzumab-dttb; Trastuzumab-pkrb; Trastuzumab-qyyp; Trazimera
Biological: Trastuzumab Emtansine — Given intravenously (IV)
  Other Names: Ado Trastuzumab Emtansine; ADO-Trastuzumab Emtansine; Kadcyla; PRO132365; RO5304020; T-DM1; Trastuzumab-DM1; Trastuzumab-MCC-DM1; Trastuzumab-MCC-DM1 Antibody-Drug Conjugate; Trastuzumab-MCC-DM1 Immunoconjugate
Drug: Vemurafenib — Given PO
  Other Names: BRAF (V600E) kinase inhibitor RO5185426; BRAF(V600E) Kinase Inhibitor RO5185426; PLX-4032; PLX4032; RG 7204; RG7204; RO 5185426; Zelboraf
Drug: Vinorelbine — Given IV
  Other Names: Dihydroxydeoxynorvinkaleukoblastine
Drug: Vismodegib — Given PO
  Other Names: Erivedge; GDC-0449; Hedgehog Antagonist GDC-0449

SUMMARY:
SMMART-ACT is a feasibility pilot study to determine if testing samples from a participant's cancer using a precision medicine approach can be used to identify specific drugs or drug combinations that can help control their disease. The safety and tolerability of the drug or drug combination is also to be studied. Another purpose is for researchers to study tumor cells to try to learn why some people respond to a certain therapy and others do not, and why some cancer drugs stop working. The study population will include participants with advanced breast, ovarian, prostate, or pancreatic malignancies, or sarcomas.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. Feasibility of utilizing a SMMART-ACT Tumor Board to select personalized advanced cancer treatment plans based on a pre-determined set of drug agents with recommended phase 2 doses (RP2Ds).

SECONDARY OBJECTIVES:

I. Safety and tolerability of assigned ACT intervention per cancer type; II. Preliminary indications of efficacy based on disease-specific responses; and.

III. Estimated survival benefit per cancer type.

EXPLORATORY OBJECTIVES:

I. Durability of a response compared to the most recent therapy on which progression occurred.

II. Changes in ability to conduct activities of daily living (ADL). III. Changes in quality of life (QOL).

IV. Feasibility of SMMART centric assessments of ongoing responses to treatment to identify mechanisms of therapy induced change, per investigator discretion. Such mechanisms may include, but will not be limited to, the following:

IVa. Changes in tumor and tumor ecosystem biology; IVb. Response and resistance to therapy.

OUTLINE:

PRE-SCREENING: Participants undergo a screening biopsy and blood collection for review and assessment of their tumor, utilizing one or more of the SMMART-Clinical Analytics Platform (SMMART-CAP) assays. The clinical assays may be used to provide an optimal and individualized treatment approach which may or may not include a SMMART-ACT treatment regimen.

SMMART-ACT TREATMENT: Prior to enrollment, participants must receive a treatment recommendation, via a SMMART-ACT Tumor Board, that consists of one or more of the pre-defined SMMART-ACT treatment regimen options. Participants are considered enrolled in SMMART-ACT if they receive a targeted SMMART-ACT treatment regimen, which may be administered in monotherapy or in combination with other targeted agents or immunotherapies, chemotherapies, or radiation. A combination treatment plan may include a two-week monotherapy lead-in, followed by a combination treatment regimen. Regardless of overall recommended treatment plan details, each SMMART-ACT study intervention must have an established RP2D that was determined in a prior clinical trial. All participants are required to undergo an On-Treatment Biopsy after two weeks on the first dose of study drug(s), and before starting Cycle 2, regardless of whether the participant is on a monotherapy, monotherapy-induction or combination regimen. Participants will continue to receive the study agent(s) after their On-Treatment Biopsy according to the biopsy results and the results of ongoing safety and clinical assessments. Treatment cycles repeat every 21 to 28 days in the absence of disease progression or unacceptable toxicity. Cycles are determined based on the study agent(s). Upon disease progression, participants are given the option to undergo an additional repeat biopsy.

Participants completing study treatment due to disease progression are followed every 3 months for 1 year, then every 6 months for 5 years. Participants completing study treatment without disease progression are followed every 6-12 weeks for up to 5 years or until disease progression, start of a new therapy, withdrawal from the study, or death, whichever occurs first.

ELIGIBILITY:
Inclusion Criteria:

* PRE-SCREENING: Written informed consent prior to any pre-screening activities, study-specific procedures or interventions.
* PRE-SCREENING: At least 18 years of age at time of informed consent. Persons of all gender identities, biological sexes, races, and ethnicities will be included.
* PRE-SCREENING: A diagnosis of advanced sarcoma or advanced prostate, breast, ovarian, or pancreatic cancer. Change in an individual's cancer can be tracked objectively according to the Prostate Cancer Working Group 3 (PCWG3) criteria for prostate cancer, and Response Evaluation Criteria in Solid Tumors version 1.1 (RECIST v1.1) criteria for sarcomas and breast, ovarian, and pancreatic cancers.
* PRE-SCREENING: Biospecimen collection, as per institutional standards, must be consented to and collection must be feasible, with the following exceptions for tissue collections:

  * Individuals with a prior successful SMMART-CAP tumor tissue sample collected within the last 90 days may be eligible, given that =<1 treatment has been received within =< 90 days of that biopsy.
* PRE-SCREENING: Eastern Cooperative Oncology Group (ECOG) performance status of =< 2.
* PRE-SCREENING: Physician assessed life expectancy of >= 6 months.
* PRIMARY TREATMENT: Documented progression after at least 1 line of prior therapy for advanced disease. If recurrence occurred within 6 months of the last dose of an adjuvant/neoadjuvant therapy, that adjuvant/neoadjuvant therapy will count as 1 line of therapy.
* PRIMARY TREATMENT: SMMART-ACT Tumor Board treatment recommendation of at least one per protocol ACT intervention based on the board's review of SMMART-CAP results on a pre-screening biopsy.
* PRIMARY TREATMENT: Absolute neutrophil count (ANC) >= 1,500 / uL (1.5 K/cu mm) (assessed at primary [post pre-screening] screening, or by the time that study intervention commences)

  * May be waived, per principal investigator (PI), on a case-by-case basis for participant populations recognized to have normal baseline values below this level
* PRIMARY TREATMENT: Platelets >= 100,000 / uL (100 K/cu mm) (assessed at primary [post pre-screening] screening, or by the time that study intervention commences)
* PRIMARY TREATMENT: Hemoglobin >= 9 g/dL (or >= 5.6 mmol/L) (assessed at primary [post pre-screening] screening, or by the time that study intervention commences)
* PRIMARY TREATMENT: Creatinine =< 1.5 x institutional upper limit of normal (IULN) OR measured or calculated creatinine clearance (glomerular filtration rate [GFR] can also be used in place of creatinine or creatinine clearance [CrCl]) >= 50 mL/min/1.73m^2. (assessed at primary [post pre-screening] screening, or by the time that study intervention commences)

  * Creatinine clearance should be calculated per institutional standard. For participants with a baseline calculated creatinine clearance below normal institutional laboratory values, a measured baseline creatinine clearance should be determined. Individuals with higher values felt to be consistent with inborn errors of metabolism will be considered on a case-by-case basis.
* PRIMARY TREATMENT: Total bilirubin =< 1.5 x IULN OR direct bilirubin IULN for individuals with total bilirubin levels > 1.5 x IULN. (assessed at primary [post pre-screening] screening, or by the time that study intervention commences)
* PRIMARY TREATMENT: Aspartate aminotransferase (AST) (serum glutamic-oxaloacetic transaminase [SGOT]) / alanine aminotransferase (ALT) (serum glutamate pyruvate transaminase [SGPT]) =< 3 x IULN. (assessed at primary [post pre-screening] screening, or by the time that study intervention commences)
* PRIMARY TREATMENT: International normalized ratio (INR) or prothrombin time (PT) =< 1.5 x upper limit of normal (ULN) unless individual is receiving anticoagulant therapy as long as PT or partial thromboplastin time (PTT) is within intended therapeutic range of intended anticoagulant therapy. (assessed at primary [post pre-screening] screening, or by the time that study intervention commences)
* PRIMARY TREATMENT: Activated partial thromboplastin time (aPTT) or PTT =< 1.5 x ULN unless participant is receiving anticoagulant therapy, as long as PT or PTT is within therapeutic range of intended anticoagulant therapy. (assessed at primary [post pre-screening] screening, or by the time that study intervention commences)
* PRIMARY TREATMENT: Body mass index (BMI) >16.0 and < 35.0 kg/m^2

  * Participants with a BMI of >= 30.0 will use ideal body weight indices in calculating the delivery of agents that are dosed based upon body surface area (i.e., mg agent/meter squared) or weight (i.e., mg agent/kg body weight)
* PRIMARY TREATMENT: Toxicities due to prior therapies should be resolved to baseline or grade 1 (per Common Terminology Criteria for Adverse Events [CTCAE] v5.0) before administration of study intervention. The following exceptions are permitted:

  * Alopecia, fatigue, and lymphopenia due to prior therapies.
  * Toxicities attributed to prior anti-cancer therapy that are not expected to resolve and to result in long lasting sequelae, (e.g., neuropathy after platinum-based therapy), may be permitted.
* PRIMARY TREATMENT: Palliative radiation therapy completed >= two weeks prior to start of SMMART-ACT treatment to a measurable disease lesion (s).
* PRIMARY TREATMENT: Additional eligibility criteria for the intended recommended therapy must also be met.
* PRIMARY TREATMENT: Study intervention-specific eligibility criteria for the intended, recommended therapy must also be met.
* CANCER SPECIFIC BREAST CANCER: Lesion(s) remain measurable after systemic therapies, as follows:

  * At least one prior line of pharmacological therapy for hormone receptor (HR) positive, human epidermal growth factor receptor 2 (HER2)-negative disease.
  * At least one prior line of targeted therapy for HER2-postive disease.
  * At least one prior line of combination therapy for triple negative disease lacking a BRCA1/2 mutation.
  * At least one prior line of therapy with a PARP inhibitor for triple negative disease with a BRCA1/2 mutation.

Exclusion Criteria:

* PRE-SCREENING: Evidence of active malignancy of another cancer with a natural or treatment history that may affect safety or efficacy assessments of this study or impose unacceptable risk to the participant. Guiding examples for those who can be enrolled include: individuals who have been disease free for two years; cancers with high cure rates (e.g., prior history of stage 1 rectal cancer and currently otherwise disease free); adequately treated localized non-melanomatous skin cancer.
* PRE-SCREENING: Involuntarily incarceration, including, but not limited to, imprisonment and compulsory detained for treatment of psychiatric or physical (e.g., infectious disease) illness.
* PRIMARY TREATMENT: Any brain/central nervous system (CNS) metastases or brain/CNS metastases that has progressed (e.g., evidence of new or enlarging brain metastasis that progresses within =< four weeks of CNS directed treatment as ascertained by clinical examination(s) and magnetic resonance imaging (MRI) or computed tomography (CT) during the main eligibility screening period.
* PRIMARY TREATMENT: One or more new, active brain/CNS metastasis or the presence of known leptomeningeal disease (LMD) that requires immediate treatment. If treatment within the first cycle of therapy is unlikely to be required, enrollment may be considered, as per the investigator.
* PRIMARY TREATMENT: Concurrent forms of anti-cancer therapy that have the potential to interfere with efficacy and safety assessments or may that may pose increased risk to the participant while on a SMMART-ACT treatment, and as per the investigator. (Select hormone therapies, are allowed.)
* PRIMARY TREATMENT: Untreated and/or uncured hepatitis C virus (HCV) infection, as evidenced by detectable hepatitis B virus (HBC) ribonucleic acid (RNA) by polymerase chain reaction (PCR). Prior treatment, concurrent treatment, and natural resolution of HCV infection are not exclusionary given (1) no risk for hepatic decompensation and (2) the intended SMMART ACT treatment is not expected to exacerbate HCV infection.
* PRIMARY TREATMENT: Uncontrolled intercurrent illness and infection that may interfere with planned treatment including, but not limited to the following:

  * Symptomatic congestive heart failure (New York Heart Association [NYHA] class III or IV)
  * Unstable angina pectoris or coronary angioplasty, or stenting within < six months prior to enrollment,
  * Cardiac arrhythmia (ongoing cardiac dysrhythmias of grade >=2 [National Cancer Institute (NCI) CTCAE v5.0]),
  * Conditions that require intra-cardiac defibrillators,
  * Known cardiac metastases,
  * History of abnormal cardiac valve morphology (>= grade 2),
  * Chronic graft versus host disease (GVHD) or immunosuppressive therapy for the control of GVHD.
* PRIMARY TREATMENT: Severe infection within < four weeks prior to initiation of study treatment, including, but not limited to, hospitalization for complications of infection, bacteremia, or severe pneumonia.
* PRIMARY TREATMENT: Inability or unwillingness to take oral medication (only for assigned oral study interventions).
* PRIMARY TREATMENT: History of allergy to an assigned study agent or its excipients.
* PRIMARY TREATMENT: Current pregnancy, currently breast-feeding, or unwillingness to not breastfeed while receiving study drug(s) or for the minimum required time after the last dose of study drug(s) as specified by the SMMART-ACT drug agents.
* PRIMARY TREATMENT: Any condition that, in the opinion of the investigator, could jeopardize the participant's safety or adherence to the study protocol.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2023-01-30 (Estimated); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of participants who receive an ACT therapy based an ACT Tumor Board recommendation. | From time of SMMART-ACT Tumor Board review to first dose of SMMART-ACT study drug regime as evaluated at interim analysis (approximately 2 years)
  At interim analysis, if greater than or equal to 11 of the first 15 enrolled participants (80%) receive C1D1 of the recommended ACT drug regimen, the feasibility threshold will be met. If not attained, reasons as to why the feasibility endpoint was not met will be reviewed.

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events | First dose of study drug up to 30 days after last dose study drug(s)
  Measured by Common Terminology Criteria for Adverse Events version 5.0.
Rate of treatment discontinuation due to toxicities and/or intolerability. | First dose of study drug to last dose study drug(s)
  Measured by Common Terminology Criteria for Adverse Events version 5.0.
Overall response rate (ORR) | At 6 months from cycle 1 day 1 +/- 2 weeks (each cycle may be 21 or 28 days, depending on the assigned SMMART ACT regimen)
  Will be assessed by ORR = complete response (CR)+ partial response (PR) per Response Evaluation Criteria in Solid Tumours (RECIST) 1.1 or in accordance with definition for pseudoprogression indications for immuno monotherapy regimens. Will be estimated using the Kaplan-Meier method.
Progression free survival | From the first dose of study drug until the earliest date of disease progression, as measured by investigator assessment, or death due to any cause (until the end of long-term follow-up (LTFU)), LTFU is up to 5 years
  Will be censored at the date of last adequate assessment visit and will be estimated using the Kaplan Meier method.
Disease-specific survival | Time from the first day of treatment with study intervention to death as a result of the disease at time of last follow-up, LTFU is up to five years from time of last dose of study therapy
  Will be estimated using cumulative incidence methods.
Overall survival | From the time of first dose of study drug until death from any cause (until the end of long-term follow-up), LTFU is up to 5 years
  Will be censored on the last date a participant is known to be alive and will summarized descriptively using the Kaplan-Meier method. The median and 95% confidence interval, will be included in the estimations, if possible.

CONTACTS AND LOCATIONS:
Overall Officials: Lara Davis, Principal Investigator — OHSU Knight Cancer Institute